CLINICAL TRIAL: NCT03617952
Title: Prices, Peers, and Perceptions: Field Experiments on Technology Adoption in the Context of Improved Cookstoves
Brief Title: P3 Ghana Cookstove Study
Acronym: P3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Colorado, Boulder (Other); North Carolina State University (Other); Navrongo Health Research Centre, Ghana (Other); U.S. National Science Foundation (U.S. Federal Agency); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-0359; SES 1528811 (Other Grant/Funding Number: NSF)
Record Dates: First submitted 2018-07-03; First posted 2018-08-07 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Household Air Pollution; Behavior, Social
Keywords: Cookstoves; Household Air Pollution; Behavior Change; Global Health
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S1 (Peer) group (Experimental): S1 group households located in 25 clusters that were included in a prior cookstove study: selected households are nearest neighbors (peers) of households who received free stoves in that prior study. This group is used to represent a potentially high peer influence on the adoption of improved cookstoves.
  The P3 Bio Intervention is implemented in this group.
  Interventions: Behavioral: P3 Bio Intervention
- S2 (Non-Peer) Group (Experimental): S2 group households are located in 25 clusters randomly selected from the area of the K-N Districts more than 1 km from the S1 clusters. This group will have minimal prior knowledge of the cookstoves through peers.
  The P3 Bio Intervention is implemented in this group.
  Interventions: Behavioral: P3 Bio Intervention

INTERVENTIONS:
Behavioral: P3 Bio Intervention — Two types of improved biomass burning cookstoves (ACE1 and Greenway Jumbo) are offered to participants in both arms at varying prices.

SUMMARY:
Background:

Despite their potential health and social benefits, adoption and use of improved cookstoves has been low throughout much of the world. Explanations for low adoption rates of these technologies include prices that are not affordable for the target populations, limited opportunities for households to learn about cookstoves through peers, and perceptions that these technologies are not appropriate for local cooking needs. The P3 project employs a novel experimental design to explore each of these factors and their interactive effects on cookstove demand, adoption, use and exposure outcomes.

Methods:

The P3 study is being conducted in the Kassena-Nankana Districts of Northern Ghana. Leveraging an earlier improved cookstove study that was conducted in this area, the central design of the P3 biomass stove experiment involves offering stoves at randomly varying prices to peers and non-peers of households that had previously received stoves for free. Using household surveys, electronic stove use monitors, and low-cost, portable monitoring equipment, we measure how prices and peers' experience affect perceptions of stove quality, the decision to purchase a stove, use of improved and traditional stoves over time, and personal exposure to air pollutants from the stoves.

Discussion:

The challenges that public health and development communities have faced in spreading adoption of potentially welfare-enhancing technologies, like improved cookstoves, have highlighted the need for interdisciplinary, multisectoral approaches. The design of the P3 project draws on economic theory, public health practice, engineering, and environmental sciences, to more fully grasp the drivers and barriers to expanding access to and uptake of cleaner stoves. Our partnership between academic institutions, in the US and Ghana, and a local environmental non-governmental organization creates unique opportunities to disseminate and scale up lessons learned.

ELIGIBILITY:
Inclusion Criteria:

* Classified as "rural"
* Uses biofuel as main cooking fuel source
* Has women in household aged 18-55 and at least one child under five

Exclusion Criteria:

* Clusters that are close to the S1 clusters, creating a set of clusters far enough from the original R group that will create the S2 cluster.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Stove Purchases | Number of households that order stoves and complete payments | up to 13 months
  Number of households in each arm that place orders for and subsequently complete all payments on the two types of stoves.

SECONDARY OUTCOMES:
Cooking Behaviors | Household use of both traditional and improved cookstoves over time | up to 13 months
  Use of traditional and improved stoves over time across intervention arms.
Perceptions of Stove Quality | Smoke production, efficiency, ease of use, quality of food, etc. | up to 13 months
  Likert-scale and subjective expectation questions measuring perceptions of stove quality / performance for both stove types along multiple dimensions. Example scale question: "How much smoke do you think the ACE1 stove would produce?" Response options: 1 = A lot less smoke than a 3 stone fire, 2 = A little less smoke than a 3 stone fire; 3 = About the same amount of smoke as a 3 stone fire; 4 = A little more smoke than a 3 stone fire; 5 = A lot more smoke than a 3 stone fire; 99 = Don't know / not sure.
Exposure to CO and PM 2.5 | up to 13 months
  Kitchen concentrations of and personal exposure to carbon monoxide (CO) and particular matter (PM2.5) among study participants

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Dickinson, PhD, Principal Investigator — Unviersity of Colorado, Aurora

IPD SHARING:
Plan to Share IPD: Yes
Survey Data; Personal exposure, proximity, and air quality data; and short term stove use and proximity data will have team access only to full data set with identifiers. De-identified data will be open access with registration and a statement of interest. Stove use data will be open access with registration and a statement of interest.
Supporting Information: Study Protocol, ICF
Time Frame: The results will be submitted for publication immediately after a sufficient level of analytical detail has been achieved through experiments and data analysis.
Access Criteria: No fee will be charged for access to the data other than applicable publication subscription fees charged by peer-reviewed journals or proceedings copy fees charged by conferences. The data will be open to wider use at the time of publication.

REFERENCES:
- [Derived] Dickinson KL, Dalaba M, Brown ZS, Alirigia R, Coffey ER, Mesenbring E, Achazanaga M, Agao D, Ali M, Kanyomse E, Awaregya J, Adagenera CA, Aburiya JBA, Gubilla B, Oduro AR, Hannigan MP. Prices, peers, and perceptions (P3): study protocol for improved biomass cookstove project in northern Ghana. BMC Public Health. 2018 Oct 29;18(1):1209. doi: 10.1186/s12889-018-6116-z. PMID 30373560

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/52/NCT03617952/Prot_SAP_000.pdf